CLINICAL TRIAL: NCT05840042
Title: Epidemiology and Risk Factors of Uterine Fibroids in China
Status: Not yet recruiting | Type: Observational
Sponsor: Shixuan Wang (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); Tongji Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); West China Hospital (Other); The Fourth Hospital of Shijiazhuang (Other)
Responsible Party: Sponsor-Investigator, Shixuan Wang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: V2.0
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Uterine fibroids are the most common form of benign uterine tumors in the uterine muscle layer, which had a certain rate of malignancy, but it is rare. The prevalence of uterine fibroids estimates range from 4.5% to 68.6% depending on study population and diagnostic methodology. The prevalence of fibroids has been historically underestimated by epidemiologic studies which focused mainly on symptomatic women, leaving behind a large population of asymptomatic women and women who underreport their symptoms. What investigators don't know was which women who have fibroids will develop clinical symptoms and which women who have an operation of myomectomy will relapse. The purpose of this study is to investigate the prevalence, incidence and risk factors for the development of uterine fibroids in Chinese women.

ELIGIBILITY:
Inclusion Criteria:

* Current place of residence≥ 6 months;
* No serious mental illness or mental abnormality;
* Those who agree to participate in this survey and cooperate in completing the questionnaire.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study population is women aged more than 18yrs with or without uterine fibroids from five regions of China. The study time period will conduct from May 1, 2023 - November 30, 2025 to allow for 6 months pre-index for evaluating baseline demographic and clinical characteristics and 24 months post-index, ensuring a minimum of one years follow-up.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-06-19 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of uterine fibroids in China | Baseline
  Prevalence of uterine fibroids in China

SECONDARY OUTCOMES:
Incidence of uterine fibroids in China | Two follow-ups over a three-year period
  Incidence of uterine fibroids in China
Risk factors of development of uterine fibroids in China | Two follow-ups over a three-year period
  Associated risk factors for recurrence, infertility and malignancy of uterine fibroids in China

CONTACTS AND LOCATIONS:
Overall Officials: SHIXUAN WANG, DOCTOR, Principal Investigator — Huazhong University of Science and Technology

REFERENCES:
- [Derived] Yan W, Yuan S, Zhou D, Zhang M, Yang S, Wang W, Wang S. Status and treatment of patients with uterine fibroids in hospitals in central China: a retrospective study from 2018 to 2021. BMJ Open. 2024 Jan 17;14(1):e081736. doi: 10.1136/bmjopen-2023-081736. PMID 38233053